CLINICAL TRIAL: NCT00005031
Title: A Phase II Evaluation of MGI-114 in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Irofulven in Treating Patients With Persistent or Recurrent, Refractory Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067554; GOG-129L
Record Dates: First submitted 2000-04-06; First posted 2004-03-31 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2008-03

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients who have persistent or recurrent refractory endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity of 6-hydroxymethylacylfulvene in patients with persistent or recurrent, refractory endometrial carcinoma. II. Determine the nature and degree of toxicity of this treatment in these patients.

OUTLINE: This is a multicenter study. Patients receive 6-hydroxymethylacylfulvene IV over 5 minutes on days 1-4. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 19-51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed endometrial carcinoma refractory to curative therapy or established treatments Clinically or histologically confirmed persistent or recurrent disease Bidimensionally measurable disease (ascites or pleural effusions not considered measurable) Not eligible for higher priority GOG protocol

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Platelet count at least 100,000/mm3 Absolute neutrophil count at least 1,500/mm3 Hepatic: Bilirubin normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No clinically uncontrolled dysrhythmia or signs of ischemia per ECG No congestive heart failure requiring medication No uncontrolled hypertension Other: No significant active infection No other prior or concurrent malignancy within the past 5 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy and recovered No more than 1 prior chemotherapy regimen allowed (either single or combination cytotoxic drug therapy) No prior 6-hydroxymethylacylfulvene No prior chemotherapy for other malignancy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No prior radiotherapy for other malignancy Surgery: At least 3 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell J. Schilder, MD, Study Chair — Fox Chase Cancer Center
Locations (40):
- United States (39):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Schilder RJ, Blessing JA, Pearl ML, Rose PG. Evaluation of irofulven (MGI-114) in the treatment of recurrent or persistent endometrial carcinoma: A phase II study of the Gynecologic Oncology Group. Invest New Drugs. 2004 Aug;22(3):343-9. doi: 10.1023/B:DRUG.0000026262.77502.31. PMID 15122083